CLINICAL TRIAL: NCT05086770
Title: Comparison of Pain After Uterine Artery Embolization Using Gelatin Microsphere or Tris-acryl Gelatin Microsphere in Patients With Symptomatic Fibroids: A Prospective, Randomized Study
Brief Title: Comparison of Pain After Uterine Artery Embolization Using Gelatin Microsphere or Tris-acryl Gelatin Microsphere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEXTBIO-UIGB-UF01
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Uterine Myoma; Uterine Fibroid
MeSH Terms: conditions — Myofibroma; Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The test group will be administered 300-500 ㎛ range of Gelatin microsphere (Nexsphere™). A suspension in which a contrast medium and physiological saline are mixed will be administered until the embolization is sufficiently achieved.
  Interventions: Device: Gelatin microsphere (Nexsphere™)
- Control group (Active Comparator): The control group will be administered 500-700 ㎛ of Embospheres until sufficient embolization is achieved.
  Interventions: Device: Embosphere

INTERVENTIONS:
Device: Gelatin microsphere (Nexsphere™) — Gelatin microsphere (Nexsphere™) is a yellow powder, made of 100% hydrophilic gelatin. It is used to make a suspension by mixing a contrast agent and physiological saline. The indications for gelatin microsphere are hepatic artery chemoembolization, uterine artery embolization, prostate artery embolization, and treatment of various hemorrhagic diseases. It physically embolizes blood vessels and is decomposed within 4-8 weeks after intravascular injection.
  Arms: Test group
Device: Embosphere — Tris-acryl gelatin microspheres (Embosphere Microspheres) are biocompatible and nonresorbable with cell adhesion properties for complete and durable mechanical occlusion.
  Arms: Control group

SUMMARY:
This study is a prospective and randomized investigation planned to compare pain after uterine artery embolization using Gelatin microsphere or tris-acryl gelatin microsphere in 60 patients with symptomatic fibroids.

DETAILED DESCRIPTION:
This investigational study is designed to compare pain after uterine artery embolization using Gelatin microsphere or tris-acryl gelatin microsphere in patients with symptomatic fibroids.

The primary end-points will be evaluated by assessing the maximum Visual Analogue Scale (VAS) score obtained for each time points within 24 hours after embolization.

Secondary end-points consist of evaluating six items: 1) fentanyl and analgesic usage within 24 hours, 2) comparison of symptom severity score and health-related quality of life score, 3) comparison of postoperative inflammation, 4) assessment of tumor necrosis degree in Magnetic Resonance Imaging, 5) fluoroscopy and procedure time comparison, and 6) assessment of residual ovarian function before and after surgery (Serum AMH).

This study included patients between the ages of 20 and less than 60 years of age who were diagnosed with uterine myoma and planned to undergo uterine artery embolization.

ELIGIBILITY:
Inclusion Criteria:

* A patient aged between 20 and under 60 who decided to undergo uterine artery embolization for symptomatic uterine myoma.

Exclusion Criteria:

* Bradycardia on electrocardiogram (< 45 bpm)
* Ventricular conduction abnormalities
* Liver failure
* Kidney failure
* Uncontrolled high blood pressure
* Obesity (BMI ≥ 30 ㎏/㎡)
* Patients who are allergic to drugs
* Patients who cannot read consent forms such as illiterate or foreigners
* Pregnant woman

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity by numerical rating scale | 0-24 hours after embolization
  0-10 numerical rating scale (0, no pain at all; 10, worst pain imaginable

SECONDARY OUTCOMES:
Fentanyl and analgesic usage volume | 24 hours
  Fentanyl and analgesic usage volume within 24 hours after embolization
Symptom severity score | 3 months
  Comparison of symptom severity score before and 3 months after embolization
  Symptom was scored on a scale of 0-10, with 0 being no symptoms and 10 being the baseline, or initial symptoms.
Postoperative inflammation | 24 hours
  Comparison of level or counts of C-Reactive Protein (CRP), leukocyte, neutrophil before and after embolization
Tumor necrosis degree | 3 months
  Assessment of tumor necrosis degree in MR after embolization
Fluoroscopy and procedure time | procedure time
  Fluoroscopy and procedure time taken for embolization to achieved
Serum Anti-Mullerian Hormone (AMH) | 3 months
  Residual ovarian function before and after embolization

CONTACTS AND LOCATIONS:
Overall Officials: Man Deuk Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea